CLINICAL TRIAL: NCT03165318
Title: A Randomized, Sham-Controlled Pilot Study of Pulsed Electromagnetic Field Therapy in Promoting the Maintenance of Muscle Following Anterior Cruciate Ligament (ACL) Reconstruction
Brief Title: Pulsed Electromagnetic Field (PEMF) Systems to Promote the Maintenance of Bone and Muscle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015/00276
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Muscle Loss Post Anterior Cruciate Ligament Reconstruction
Keywords: Pulsed electromagnetic field; Anterior cruciate ligament reconstruction; Muscle

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed Electromagnetic Field Therapy (Active Comparator): Active Pulsed Electromagnetic Field therapy device; exposed once weekly for 10 minutes.
  Interventions: Device: Pulsed Electromagnetic Field Therapy
- Sham Therapy (Sham Comparator): Inactive Pulsed Electromagnetic Field therapy device; exposed once weekly for 10 minutes.
  Interventions: Device: Sham Therapy

INTERVENTIONS:
Device: Pulsed Electromagnetic Field Therapy — Participants of this arm will be exposed to 10 minutes of Pulsed Electromagnetic Field (PEMF) once a week for a total of 16 weeks.
  The PEMF device produces pulsed magnetic fields at flux densities up to 1 mT peak.
  Arms: Pulsed Electromagnetic Field Therapy
Device: Sham Therapy — Participants of this arm will be exposed to 10 minutes of sham therapy once a week for a total of 16 weeks.
  The Sham device is identical to the PEMF device in physical appearance.
  Arms: Sham Therapy

SUMMARY:
This is a pilot study that evaluates the effect of PEMF in maintaining muscle mass postoperatively in individuals experiencing clinical immobilisation due ACL reconstruction surgery. Half of the participants will receive the PEMF therapy in combination with standard rehabilitation programme, while the other half will receive sham therapy in combination with standard rehabilitation programme.

DETAILED DESCRIPTION:
This is a single-site, randomized, double-blinded, prospective pilot study of the effectiveness of once-weekly PEMF therapy in the promotion of muscle maintenance following ACL reconstruction surgery. Eligible subjects will be randomized in a 1:1 ratio to receive therapy with an active PEMF device or an identical inactive Sham device, in addition to the standard rehabilitation regimen.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have undergone unilateral first-time athroscopic reconstruction with single bundle hamstring graft using both transtibial and transportal techniques for rupture anterior cruciate ligament
* Informed consent signed

Exclusion Criteria:

* Subjects requiring concomitant knee ligament reconstruction
* Subjects having other than hamstring graft for the ACL reconstruction
* Subjects with history of cardiac, neurological, and rheumatological diseases, and previous lower limb surgery/ fracture
* Subjects with Leg circumference > 63 cm
* Pregnant women

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2017-03-07 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Muscle Volume | Week 1 and Week 16 post-ACL reconstruction
  % change in muscle volume at the end of 16 weeks compared to baseline

SECONDARY OUTCOMES:
Quadriceps strength | Baseline and Week 8, 12, 16 post-ACL reconstruction
  Quadricep strength (Ib) measurement by dynamometer
Knee and thigh circumference | Baseline and Week 1, 4, 8, 12, 16 post-ACL reconstruction
  Measurement of knee girth (cm) from mid portion of the patella and thigh girth (cm) 5 cm above from the superior border of the patella
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Week 16 post-ACL reconstruction
  Knee Injury and Osteoarthritis Outcome Score (KOOS): a validated knee-specific instrument that measures the short-term and long-term symptoms and function associated with knee injury. KOOS consists of 5 subscales: pain, other symptoms, function in daily living, function in sport and recreation, and knee related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Lingaraj Krishna, frcs (Orth), Principal Investigator — National University Health System
Locations (1):
- National University Health System, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No